CLINICAL TRIAL: NCT03620591
Title: Intraoperative Use of Lidocaine and Postoperative Analgesia After Laparoscopic Cholecystectomy
Brief Title: Lidocaine and Analgesia After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Baloyiannis, Assistant Professor of Surgery, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UHL27823/06/28/2018
Record Dates: First submitted 2018-07-18; First posted 2018-08-08 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain; Opioid Consumption
Keywords: Lidocaine; Postoperative Pain; Opioid consumption; Laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Intraoperative administration of lidocaine to patients undergo laparoscopic cholecystectomy.
  Prior induction to anesthesia, lidocaine bolus 1.5 mg / kg will be administered to the lidocaine group and then patients will be connected to a continuous 2 mg / kg / h administration of lidocaine until the end of the procedure.
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Intraoperative administration of normal saline to patients undergo laparoscopic cholecystectomy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Intraoperative administration of lidocaine
  Arms: Lidocaine
Drug: Placebo — Intraoperative administration of normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how effective is the intraoperative use of lidocaine to attenuate postoperative pain and opioids consumption after laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Acute postoperative pain may predict the development of chronic pain.Recently, the analgesic effect of lidocaine, as a part of a multimodal analgesia, has been evaluated in many studies. They have shown that lidocaine may have a role in the postoperative pain management, as an adjunct.

Acute postoperative pain after laparoscopic cholecystectomy is complex in nature. Postoperative pain is the main complaint and the primary reason for delay discharge after laparoscopic cholecystectomy.The study includes patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Age ≥ 18 years old
* BMI ≤ 35

Exclusion Criteria:

* Allergy in local anesthetics
* History of liver, kidney or heart failure
* Existence of chronic pain history or daily analgesics
* Psychiatric disorders
* Inability to understand pain assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours after the procedure
  The total dose of tramadol is calculated as mg and administered intravenously.

SECONDARY OUTCOMES:
Postoperative pain | Departure of the patient from the recovery room (0hrs)
  Numeric Rate scale 0-10 (0=no pain to 10=worst imaginable pain)
Postoperative pain | 6 hrs after the procedure
  Numeric Rate scale 0-10 (0=no pain to 10=worst imaginable pain)
Postoperative pain | 12 hrs after the procedure
  Numeric Rate scale 0-10 (0=no pain to 10=worst imaginable pain)
Postoperative pain | 24 hrs after the procedure
  Numeric Rate scale 0-10 (0=no pain to 10=worst imaginable pain)
Incidence of Nausea and Vomiting | 24 hours
  The percentage of patients who had nausea and vomiting during the first 24 hours
Incidence of sedation and respiratory depression | 24 hours
  The percentage of patients who had sedation and respiratory depression during the first 24 hours
Incidence of shoulder pain | 24 hours
  The percentage of patients who had shoulder pain during the first24 hours
Incidence of headache and dizziness | 24 hours
  The percentage of patients who had headache and dizziness during the first 24 hours
Change from baseline Mean Blood Pressure | Intraoperative
  Non-invasive blood pressure measurement by using sphygmomanometer cuff
Change from Baseline Heart Rate | Intraoperative
  Bradycardia, tachycardia during the procedure
Change in depth of anesthesia | Intraoperative
  Maintenance of Bispectral index (BIS) values of 40 to 50
Side effect related to administration of lidocaine | 24 hours
  The percentage of patients who had tremor, dizziness, dysarthria, agitation, hallucinations and drowsiness during the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Baloyiannis, Study Director — University Hospital of Larissa; Chamaidi Sarakatsianou, Principal Investigator — University Hospital of Larissa; Stavroula Georgopoulou, Study Chair — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Greece